CLINICAL TRIAL: NCT03504176
Title: Pediatric Acute Respiratory Distress Syndrome Bundle vs. Standard Care; a Before-and-After Study
Brief Title: Pediatric Acute Respiratory Distress Syndrome Ventilation Bundle
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Judith Wong Ju-Ming, Dr, KK Women's and Children's Hospital
Other Study IDs: 2017/3076
Record Dates: First submitted 2018-04-08; First posted 2018-04-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Patients will be ventilated according to the bundle; including ventilation targets, tidal volume, end expiratory pressure-fraction of inspired oxygen titration.
  Interventions: Other: Ventilation bundle
- Control: Standard of care prior to implementation of the ventilation bundle

INTERVENTIONS:
Other: Ventilation bundle — ventilation targets (pH, spO2, pCO2) tidal volume 3-6ml/kg peak pressures <28-32cmH2O PEEP-FiO2 titration tables
  Groups: Intervention

SUMMARY:
Mortality rates in children with pediatric acute respiratory distress syndrome (PARDS) are higher in Asia compared to other regions. In adults with acute respiratory distress syndrome, the only therapy that improves mortality rates is a lung protective ventilation strategy. The pediatric ventilation recommendations by the Pediatric Acute Lung Injury Consensus Conference (PALICC) are extrapolated from evidence in adults, including ventilation with low tidal volume, low peak/plateau pressures and high end expiratory pressure. A recent retrospective study of ventilation practices in Asia including Singapore showed that a majority of patients with PARDS were being ventilated with high tidal volume, high peak pressure and low end expiratory pressure, not in compliance with PALICC recommendations. We postulate that currently used ventilation strategies could have contributed to the high PARDS mortality rates in Asia. We aim to determine if implementing a ventilation bundle comprising PALICC recommendations lowers PARDS and pediatric intensive care unit (PICU) mortality rates.

DETAILED DESCRIPTION:
We implement a PARDS ventilation bundle compliant with PALICC recommendations. The bundle contains a daily checklist for ventilation targets and reference tables listing targeted tidal volumes and end expiratory pressure-fraction of inspired oxygen titration. We will recruit mechanically ventilated patients who meet PARDS criteria. After a one-month implementation period, we will collect patient data over the subsequent 18 months, and compare them with the corresponding data in the 24 months prior to the implementation. The primary outcome is PARDS mortality, defined as number of deaths out of PARDS cases. Secondary outcomes are feasibility of ventilation bundle implementation, ventilator (VFD) and intensive care unit (IFD) free days and PICU mortality (number of deaths out of PICU admissions).

ELIGIBILITY:
Inclusion Criteria:

* fulfill criteria for PARDS
* mechanically ventilated

Exclusion Criteria:

* perinatal lung disease

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children admitted to the PICU needing mechanical ventilation will be screened for eligibility. Those who fulfill the PALICC criteria for PARDS will be included.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
mortality | up to 60 days
  death during PICU stay

SECONDARY OUTCOMES:
ventilator free days | up to 28 days
  days alive and free from mechanical ventilation
PICU free days | up to 28 days
  days alive and discharged from PICU

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No